CLINICAL TRIAL: NCT05839132
Title: Clinical Effect of Acupuncture in Neurodegenerative Diseases on Traumatic Brain Injury Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMUH111-REC1-239
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Neurodegenerative Diseases
Keywords: Acupuncture; Traumatic Brain Injury
MeSH Terms: conditions — Neurodegenerative Diseases; Brain Injuries, Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture treatment group (Experimental): Disposable acupuncture needles will be inserted into acupoints for a depth of 20-30 mm in a direction oblique or parallel to the surface. To ensure allocation concealment, all needles will be affixed with plastic O-rings and adhesive tapes.
  Acupuncture points: Baihui(DU20), Sishencong(EM1), Hegu(LI4), Taichong(LR3)
  Interventions: Procedure: Acupuncture
- sham acupuncture treatment group (Placebo Comparator): Streitberger's non-invasive placebo acupuncture needles will be used in the control group; blunt-tipped needles will touch the skin quickly without being inserted. To ensure allocation concealment, all needles will be affixed with plastic O-rings and adhesive tapes.
  Acupuncture points: Baihui(DU20), Sishencong(EM1), Hegu(LI4), Taichong(LR3)
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — 20 minutes of acupuncture treatment, twice a week for 2 weeks. Acupoints will be manually stimulated every 10 minutes.

SUMMARY:
Traumatic brain injury (TBI) is an altered brain function caused by an external force, which may annually have 69 million incidence cases all over the world. Increasing evidence suggests that TBI may be a major risk of beta amyloid (Aβ)-associated neurodegenerative disorders, such as Alzheimer's disease, frontotemporal dementia, and Parkinson's disease. Investigations from brain imaging studies revealed that Aβ density maps of TBI patients overlapped with those with Alzheimer's disease, and increased Aβ density not only associated with prolonged TBI duration but also associated with decreased white matter integrity. It has been suggested that the axonal injury and cerebrovascular dysfunction due to TBI may associate with the elevated level of Aβ peptides. The increasing accumulation in Aβ due to TBI may contribute to the initiation of the pathological alterations in neurodegeneration diseases. Recent animal studies suggest that acupuncture may promote regeneration of nerves in injured tissues and reduce the concentration of Aβ in brain. Moreover, recent clinical trials also indicate that acupuncture may improve the vascular cognitive impairment due to cerebral small vessel disease. Thus, acupuncture treatment on TBI may not only be of benefit for the TBI recovery but also act to interrupt the pathological changes in these neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 20 years old
2. GCS score > 8
3. loss of consciousness < 24 hr
4. the physical condition is suitable for acupuncture treatment
5. having adequate competency for understanding the study and a willingness to sign the written informed consent forms
6. be able to commence the acupuncture intervention within 2 weeks after TBI diagnosis

Exclusion Criteria:

1. medical history of neurological, cardiovascular events, e.g., epilepsy, stroke, major depression or anxiety
2. a history of the mental disorder, e.g., major depression or anxiety
3. other major medical conditions, e.g., active cancer, uncontrolled diabetes, amputation
4. receipt of acupuncture within the 6 months prior to study entry
5. patients with pacemaker or metal graf

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
plasma levels of Aβ peptide | After 2-week acupuncture treatment interva
  Decreased plasma levels of Aβ peptide
plasma levels of tau | After 2-week acupuncture treatment interva
  Decreased plasma levels of tau
plasma levels of glial fibrillary acidic protein (GFAP) | After 2-week acupuncture treatment interva
  Decreased plasma levels of glial fibrillary acidic protein (GFAP)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided